CLINICAL TRIAL: NCT04269109
Title: A Multi-modal, Opioid Sparing Pain Management Strategy in Cardiac Surgery
Brief Title: Opioid Sparing Pain Management Strategy
Status: Completed | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00085849
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Cohort: A control cohort from September 1, 2018 - October 31, 2018
  Interventions: Other: Multi-modal Opioid Sparing Pain Management Protocol
- Intervention Cohort: An intervention cohort from March 1, 2019 - April 30, 2019
  Interventions: Other: Multi-modal Opioid Sparing Pain Management Protocol

INTERVENTIONS:
Other: Multi-modal Opioid Sparing Pain Management Protocol — Incorporating multimodal opioid sparing ERAS techniques for cardiac surgery patients should show a decrease in the amount of opioids received, reduction in incidence of chronic pain, ileus, delirium, and potential for opioid addiction post-operatively. Between the dates of November 2018 through February 2019, a multi-modal, opioid sparing pain management protocol was evolving and a protocol was put into place. This study will compare outcomes before and after implementation of the protocol between the dates of September 1, 2018 - October 31, 2018 and March 1, 2019 - April 30, 2019.

SUMMARY:
The purpose of this research study is to compare the amount of morphine milligram equivalents consumed post operatively until discharge between the control cohort and intervention cohort.

DETAILED DESCRIPTION:
Retrospective data will be collected on patients admitted to Prisma Health-Upstate Greenville Memorial Hospital in the Cardiovascular Intensive Care Unit following cardiovascular surgery. They will be divided into two cohorts, a control cohort from September 1, 2018 - October 31, 2018 and an intervention cohort from March 1, 2019 - April 30, 2019. A study investigator will assess each participant's electronic medical record through the electronic medical record database - EPIC to determine eligibility per the protocol. Demographic information will be collected, including age, date of birth, race, sex, height, weight, and ethnicity. Extubation and reintubation status will be collected along with medical history, type of cardiovascular procedure, medications, length of stay, pain scores, complications, and labs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 and over
* Patients who underwent cardiac surgery requiring a coronary pulmonary bypass machine during September 1, 2018 - April 30, 2019

Exclusion Criteria:

* Patients being placed on Extracorporeal Membrane Oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This retrospective study is a self-controlled comparison of patients undergoing cardiovascular surgery by cardiovascular surgeons at Greenville Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Morphine Milligram Equivalents Comparison | 1 year
  Compare the amount of morphine milligram equivalents consumed post operatively until discharge between groups.

SECONDARY OUTCOMES:
Ileus | 1 year
  Compare incidence of postoperative ileus between both cohorts.
Delirium | 1 year
  Compare incidence of delirium between both cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline McKillop, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Prisma Health-Upstate, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Li M, Zhang J, Gan TJ, Qin G, Wang L, Zhu M, Zhang Z, Pan Y, Ye Z, Zhang F, Chen X, Lin G, Huang L, Luo W, Guo Q, Wang E. Enhanced recovery after surgery pathway for patients undergoing cardiac surgery: a randomized clinical trial. Eur J Cardiothorac Surg. 2018 Sep 1;54(3):491-497. doi: 10.1093/ejcts/ezy100. PMID 29514224